CLINICAL TRIAL: NCT07010731
Title: Level of Social Support and Associated Factors Among Diabetic Patients in Bahir Dar City Public Hospitals
Brief Title: Level of Social Support and Associated Factors Among Diabetic Patients in Bahir Dar City Public Hospitals, Amhara Regional State, North West Ethiopia, 2023
Status: Completed | Type: Observational
Sponsor: Debre Berhan University (Other)
Responsible Party: Principal Investigator, Bekalu Mekonen Belay, Mr, Debre Berhan University
Other Study IDs: BDU762/2023
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Social Support and Associated Factors Among Diabetic Patients
Keywords: social support, diabetes mellitus, family support, support system
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- After collecting the raw data and verifying its completeness, it was entered into Epi Data Software
  Interventions: Other: Social support

INTERVENTIONS:
Other: Social support — After adopting the questioner from Oslo-3 -item social support scale, it was translated in to local language (Amharic) and then back to English by another language expert. The data was collected through face-to-face interviews with three BSc nurses. It was supervised by one MSc nurse

SUMMARY:
Supplementary: English version of the questioner PART 1- Questions Related to Socio-economic Characteristics Identification No.__________________ No. Question circle the appropriate option 100 Gender of the respondent? 1. Male 2. Female 101 What is the age of the respondent? Age in years _______ (yy) 102 Residence 1. Urban 2. Rural 103 What is the educational status of the respondent? 1. no formal education 2. Grade1-8 3. Grade 9-12 4. College & above

104 monthly income of the Respondent _______ ETB 105 marital status 1. Married 2. Single 3. Widowed 4. Divorced 106 Do have health insurance 1. Yes 2. no

107 Occupation 1.Private business 2.Government employee 3.Private employee 4.other

PART 4: Clinical parameter 200 Types of diabetes 1. Type 1 2. Type 2 201 Type of current diabetic treatment 1. Insulin 2. Oral drug 3. Both 202 Duration of DM after first diagnosis. 1. < 5 years 3. >10years 2. 5-10 years 203 Comorbid status 1.Yes if specify ----------- 2.no 204 Blood glucose level 1______,2_________,3¬¬_______mg/dl

Part 3 Oslo social support scale (OSSS-3) S.no Question Response 300 How many people are so close to you that you can count on them if you have great personal problems? 1 'none' 2 '1-2' 3 '3-5' 4 '5+' 301 How much interest and concern do people show in what you do? 1 'none' 2 'little' 3 'uncertain' 4 'some' 5 'a lot' 302 How easy is it to get practical help from neighbors if you should need 1 'very difficult' 2 'difficult' 3 'possible' 4 easy 5 very easy

ELIGIBILITY:
Inclusion Criteria:The study population was a diabetic patient with a follow-up who fulfilled the eligibility criteria -

Exclusion Criteria:Those patients who are critically ill and those less than 18 years old was excluded because they couldn't provide adequate information related to the study.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adult diabetic patients were considered to be the source population
Sampling Method: Probability Sample
Enrollment: 384 (Actual)
Dates: Start 2025-04-20 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Level of social support and associated factors among diabetic patients in Bahir Dar city public hospitals, Amhara regional state, North West Ethiopia, 2023. | March 20 to April 20, 2023 GC

CONTACTS AND LOCATIONS:
Locations (1):
- Bahir Dar city public hospitals, Bahir Dar, Ethiopia

IPD SHARING:
Plan to Share IPD: Undecided